CLINICAL TRIAL: NCT00651131
Title: Cubicin(R) for Complicated Post-surgical Wound Infections
Acronym: PSW
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: terminated due to slow enrollment
Sponsor: Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3009-011; DAP-4PSW-03-03 (Other: Cubist Study Number)
Record Dates: First submitted 2008-03-31; First posted 2008-04-02 (Estimated); Last update posted 2017-08-30 (Actual); Status verified 2017-08

CONDITIONS: Wound Infections
Keywords: post-surgical; wound infection; superficial; deep; surgical
MeSH Terms: conditions — Wound Infection | interventions — Daptomycin; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: daptomycin — daptomycin i.v. 4 mg/kg q24h for 7-14 days
  Other Names: Cubicin; daptomycin for injection; Cubicin (daptomycin for injection)

SUMMARY:
The purpose of the study is to describe the clinical efficacy of CUBICIN therapy in patients with superficial and deep post-surgical Gram-positive wound infections

DETAILED DESCRIPTION:
A multi-center, single-arm, open-label, non-comparative study to describe the clinical efficacy of CUBICIN therapy in patients with superficial and deep post-surgical Gram-positive wound infections. Adjunctive treatment with aztreonam and/or metronidazole could be given for Gram-negative and/or anaerobic organisms. Patients are to be treated for a period of 7-14 days as specified in the package insert. An evaluation is to be performed on the day CUBICIN treatment is completed (assessment for outcome of cure, improved, failure or unable to evaluate). A follow-up is required for patients with an Investigator response of 'Improved' at the end of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Read and signed informed consent form
* female of childbearing potential, negative pregnancy test result
* Confirmed diagnosis of post-surgical wound infections known or suspected (based on Gram stain) to be due to Gram-positive organisms obtained within 3 calendar days prior to first dose of study medication
* Onset of surgical wound infection within 30 days after surgery
* At least three clinical signs and symptoms of skin infection

Exclusion Criteria:

* previous systemic antimicrobial therapy exceeding 24 hours duration administered anytime during 72 hours prior to the first dose of study drug
* Uncomplicated surgical infections (eg, stitch abscesses)
* osteomyelitis, pneumonia, bacteremia, endocarditis, or urinary tract infection
* Any type of space infection
* Conditions requiring surgical removal of wound infection
* necrotizing fasciitis, synergistic gangrene, Clostridial myonecrosis (gas gangrene), or Fournier's gangrene;
* Foreign material involved in the post-surgical wound infection
* Known to be allergic or intolerant to study medication
* Creatinine Clearance (CLCR) <30 mL/min
* history of neurological disease (eg, Guillain-Barré, multiple sclerosis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2004-06-01 (Actual); Primary Completion 2005-03-01 (Actual); Study Completion 2005-03-01 (Actual)

PRIMARY OUTCOMES:
Investigator's assessment of clinical response based on improvement of signs and symptoms | End of Therapy

SECONDARY OUTCOMES:
Incidence of adverse events | first dose to end of therapy
eradication of pathogens isolated at admission | End of Therapy
overall therapeutic outcome based on agreement between clinical efficacy and microbiological response | End of Therapy